CLINICAL TRIAL: NCT06888180
Title: Survey on Non-Invasive Ventilation Settings in the Intensive Care Unit for Acute Exacerbation of Chronic Obstructive Pulmonary Disease
Brief Title: Survey on NIV Settings in the Intensive Care Unit for Acute Exacerbation of COPD
Acronym: NIV-ICU
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: 2024120510170200000180001753
Record Dates: First submitted 2025-03-11; First posted 2025-03-21 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: COPD (Chronic Obstructive Pulmonary Disease); Acute Exacerbation of COPD; Hypercapnic Respiratory Failure, COPD
Keywords: COPD; Acute exacerbation of COPD; Non invasive ventilation; Hypercapnic respiratory failure
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COPD patients managed with NIV during acute exacerbation
  Interventions: Other: Non interventional study

INTERVENTIONS:
Other: Non interventional study — Documentation of Non-Invasive Ventilation Settings at Different Stages of Patient Management"

SUMMARY:
Introduction Chronic obstructive pulmonary disease (COPD) is a common condition and the fourth leading cause of death worldwide. With the rise of non-invasive ventilation (NIV), mortality among patients admitted for acute hypercapnic respiratory failure has decreased, though to a lesser extent than reported in the studies that validated this technique. We hypothesize that inappropriate initial ventilatory parameter settings for NIV could be associated with increased morbidity and mortality in this context.

Objective The primary objective of this study is to assess the initial NIV settings used in intensive care units (ICUs) and respiratory intensive care or medical intensive care units (MICUs) in this patient population. A secondary objective is to evaluate whether specific ventilatory settings are associated with mortality or the need for invasive mechanical ventilation (IMV).

Methods This is a prospective multicenter observational study aiming to include 976 patients. NIV settings will be recorded at initiation, after the first recommended arterial blood gas (ABG) evaluation (between 1.5 and 2 hours of ventilation), and at 24 and 48 hours. Patient characteristics, including medical history, clinical and biological parameters at admission, will be collected. Vital status and the need for IMV will be recorded at ICU discharge and on day 28 (D28).

ELIGIBILITY:
Inclusion Criteria:

* Adult COPD Patient
* Known or suspected COPD diagnosis as assessed by the attending physicians
* Admitted to a medical intensive care unit (MICU), respiratory intensive care unit, or MICU
* Hypercapnic respiratory distress
* NIV indication determined by the physician
* Covered by social security

Exclusion Criteria:

* Pregnant or breastfeeding women
* Other obstructive diseases (asthma, bronchiectasis, cystic fibrosis, bronchiolitis, pulmonary fibrosis, restrictive thoracic syndrome) Central hypoventilation (Ondine's syndrome, iatrogenic), neurological (neuromuscular disease), osteoarticular (kyphoscoliosis), or ENT-related causes
* Immediate need for intubation
* Acute pulmonary edema
* Contraindications to NIV (untreated pneumothorax, shock, cardiac arrest, uncontrolled vomiting, upper gastrointestinal bleeding, cervicofacial trauma, coma except when related to hypercapnia)
* Patients under legal guardianship
* Incarcerated individuals

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COPD Patients Admitted to Critical Care for Hypercapnic Respiratory Distress
Sampling Method: Non-Probability Sample
Enrollment: 976 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Ventilatory Settings at Initiation of Non-Invasive Ventilation Upon ICU Admission | Upon ICU admission

SECONDARY OUTCOMES:
Ventilatory Settings at Initiation of Non-Invasive Ventilation at 24h of ICU Admission | 24hours from ICU admission
Ventilatory Settings at 48 Hours After Initiation of Non-Invasive Ventilation in the ICU | 48hours after ICU admission
arterial blood gaz | Upon ICU admission, 24hours after ICU admission, 48hours after admission
Mortality | at 28 days

IPD SHARING:
Plan to Share IPD: Undecided